CLINICAL TRIAL: NCT01373684
Title: Induction of HBsAg Decline Using an add-on Treatment of Peginterferon Alfa-2a in HBeAg-negative Chronic Hepatitis B Patients Treated With Nucleos(t)Ide Analogous (PAS)
Brief Title: PEG-interferon Alfa-2a add-on Study in HBeAg Negative Chronic Hepatitis B Patients
Acronym: PAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBV11-01
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; HBeAg-negative
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; entecavir; Tenofovir; adefovir; adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peginterferon alfa-2a add on (Experimental): All patients are all currently being treated with long-term NA treatment. PEG-IFN will be given in a dose of 180 μg per week s.c. for a total duration of 48 weeks starting at week 0.
  Interventions: Drug: Peginterferon alfa-2a
- Nucleoside analogue (Active Comparator): All patients are all currently being treated with long-term Nucleos(t)ide analogue treatment and will continue using this medication during the duration of the study.
  Interventions: Drug: Nucleos(t)ide analogue

INTERVENTIONS:
Drug: Peginterferon alfa-2a — 180 μg per week s.c. for a total duration of 48 weeks.
  Other Names: Pegasys
  Arms: Peginterferon alfa-2a add on
Drug: Nucleos(t)ide analogue — All patients are all currently being treated with long-term NA treatment and will continue using these during the study. Dosage depends on which Nucleos(t)ide analogue they are using.
  Other Names: Entecavir (Baraclude); Tenofovir (Viread); Adefovir (Hepsera)
  Arms: Nucleoside analogue

SUMMARY:
This study intends to investigate whether addition of PEG-IFN alfa-2a in HBeAg-negative chronic hepatitis B patients who are pretreated with nucleos(t)ide analogues enhances the degree of HBsAg decline.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) is one of the most serious health problems affecting more than 350 million people worldwide, accounting for one million deaths every year. Hepatitis B e antigen (HBeAg)-negative chronic hepatitis B represents a late phase in the course of the infection, which is recognized worldwide with increasing prevalence. Therapeutic intervention is often indicated for HBeAg-negative patients because spontaneous remission rarely occurs and patients usually have more advanced liver disease in comparison with HBeAg-positive patients. With the introduction of nucleos(t)ide analogues (NA), an important progress has been made regarding antiviral therapy of CHB, but the management of the HBeAg-negative type remains difficult. NA target the reverse transcriptase of hepatitis B virus (HBV) and are potent inhibitors of viral replication. Initiation of treatment in HBeAg-negative CHB usually results in a rapid decline of serum HBV DNA levels, which is often accompanied by normalization of serum aminotransferases. However, response to treatment may not be durable in a large proportion of patients after discontinuation of therapy, indicating the necessity of long-term, and maybe indefinite, treatment. Although NA are well-tolerated during the first years of treatment, little is known about long-term safety and resistance. In contrast, the antiviral potency of peginterferon (PEG-IFN) is inferior to nucleoside analogues, but response to PEG-IFN probably is more durable in the majority of patients due to its immunomodulatory effects. Sustained off-treatment responses can be achieved in about 25% of patients treated with PEG-IFN for 1 year.

Natural killer (NK) cells are innate immune cells that not only represent the first line of defense against viral infections but play also an important role in controlling adaptive responses. The numerous mechanisms evolved by viruses to inhibit NK cell activity, as already demonstrated for HIV and HCV, may not be directed at the innate immune response, but may represent a strategy to prevent effective induction of adaptive immune responses. Defective T cell activity observed in viral infection may therefore represent a bystander effect of viral NK cell inhibition.

Recent findings of our group demonstrate that NK cells derived from the peripheral blood of chronic HBV patients display an impaired capacity to produce IFNgamma, an important cytokine for the skewing of virus-specific Th-1 responses, compared to healthy controls. Since HBV has been shown to be able to directly interfere with immune cells as well as IFNalpha-induced intracellular signalling, viral load reduction may not only improve the function of immune cells, it may also facilitate the response to PEG-IFNalpha therapy and subsequently the induction of an effective HBV-specific immune response. Treatment with a nucleoside analogue and subsequent viral decline has already shown to restore helper T-cell (TH-cell) and cytotoxic T-cell (CTL) responsiveness in chronic HBV infected patients.

Add-on treatment with PEG-IFN can be expected to further stimulate adaptive immune reactivity and may therefore result in higher rates of response.

Previous studies investigating the effect of lowering viral load with NA therapy in HBeAg-positive CHB prior to the initiation of PEG-IFN showed promising response rates to treatment. A study by Sarin et al. showed a significantly higher rate of sustained HBeAg loss in patients who received 4 weeks of lamivudine before PEG-IFN therapy (n=36) compared to those receiving placebo for 4 weeks (n=27) (36% vs. 15%, p=0.05). This treatment strategy has however not yet been applied to HBeAg-negative patients. Current guidelines recommend continuation of NA therapy for HBeAg-negative CHB until hepatitis B surface antigen (HBsAg) is cleared from serum. However, HBsAg loss rarely occurs during NA therapy in HBeAg-negative patients. In contrast, PEG-IFN therapy is associated with increasing rates of HBsAg loss every year after discontinuation of therapy.

In a study by Chan et al. HBsAg remained stable in HBeAg-positive patients and tended to reduce slowly in HBeAg-negative patients. They concluded that reduction of HBsAg for >1 log IU/mL could reflect improved immune control. It was previously shown in a study of our group that 14% of HBeAg-negative CHB patients had an HBsAg concentration decline of > 1 log after 24 weeks of therapy with PEG-IFN. Moucari et al. found an HBsAg decline of > 1 log in 25% of their patients at week 24, with mean decreases of 0.8, 1.5, and 2.1 log IU/mL at weeks 12, 24, and 48, respectively. Another study showed that 22% of patients had an HBsAg concentration decline of > 1 log after 48 weeks of treatment, which was significantly associated with HBsAg clearance three years after treatment with PEG-IFN. However, recent studies also showed that HBsAg levels do not decrease during prolonged NA therapy of HBeAg-negative CHB. Addition of PEG-IFN to NA therapy in HBeAg-negative patients may therefore be necessary to induce a decline in HBsAg levels, a first step towards subsequent HBsAg loss.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B (HBsAg positive > 6 months)
* HBeAg negative within six months prior to initiation of peginterferon alfa-2a
* HBV DNA < 200 IU/ml during nucleos(t)ide analogue (except Telbivudine) treatment within one month prior to initiation of peginterferon alfa-2a
* Compensated liver disease
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Treatment with any investigational drug within 30 days of entry to this protocol
* Current treatment with Telbivudine
* Severe hepatitis activity as documented by ALT>10 x ULN
* History of decompensated cirrhosis (defined as jaundice in the presence of cirrhosis, ascites, bleeding gastric or esophageal varices or encephalopathy)
* Pre-existent neutropenia (neutrophils <1,500/mm3) or thrombocytopenia (platelets < 90,000/mm3)
* Co-infection with hepatitis C virus, hepatitis D virus or human immunodeficiency virus (HIV)
* Other acquired or inherited causes of liver disease: alcoholic liver disease, obesity induced liver disease, drug related liver disease, auto-immune hepatitis, hemochromatosis, Wilson's disease or alpha-1 antitrypsin deficiency
* Alpha fetoprotein > 50 ng/ml
* Hyper- or hypothyroidism (subjects requiring medication to maintain TSH levels in the normal range are eligible if all other inclusion/exclusion criteria are met)
* Immune suppressive treatment within the previous 6 months
* Contra-indications for alfa-interferon therapy like suspected hypersensitivity to interferon or Peginterferon or any known pre-existing medical condition that could interfere with the patient's participation in and completion of the study.
* Pregnancy, breast-feeding
* Other significant medical illness that might interfere with this study: significant pulmonary dysfunction in the previous 6 months, malignancy other than skin basocellular carcinoma in previous 5 years, immunodeficiency syndromes (e.g. HIV positivity, auto-immune diseases, organ transplants other than cornea and hair transplant)
* Any medical condition requiring, or likely to require chronic systemic administration of steroids, during the course of the study
* Substance abuse, such as alcohol (>80 g/day), I.V. drugs and inhaled drugs in the past 2 years.
* Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-05-25 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
HBsAg decline | week 48
  HBsAg decline > 1 log from baseline at week 48

SECONDARY OUTCOMES:
HBsAg decline | week 24 and 72
  HBsAg decline > 1 log at weeks 24 and 72
HBsAg decline | week 24 and 48
  HBsAg decline > 0.5 log at weeks 24 and 48
HBsAg loss | week 48 and 72
  HBsAg loss at weeks 48 and 72

CONTACTS AND LOCATIONS:
Overall Officials: H.L.A. Janssen, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (8):
- Toronto General Hospital, Toronto, Ontario, Canada
- Netherlands (7):
  - Erasmus Medical Center, Rotterdam, South Holland
  - Onze Lieve Vrouwen Gasthuis, Amsterdam
  - VU university medical center, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Reinier de Graaf Gasthuis, Delft
  - Spaarne Gasthuis, Haarlem
  - University Medical Center Utrecht, Utrecht